CLINICAL TRIAL: NCT03555942
Title: Follicular or Luteal Start Ovarian Stimulation With Corifollitropin Alfa. A Prospective Equivalence Study With Repeated Ovarian Stimulation in Oocyte Donors
Brief Title: Luteal Phase-start Ovarian Stimulation With Corifollitropin Alfa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Nikolaos Polyzos, Clinical and Scientific Director, Fundacion Dexeus
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FSD-COR-2017-01
Record Dates: First submitted 2018-05-08; First posted 2018-06-14 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Overall, 44 oocyte donors women will be asked to participate in a trial in which they will undergo 2 consecutive ovarian stimulation protocols within a period of 6 months with 150μg corifollitropin alfa followed by 200 IU rFSH in a fixed GnRH antagonist protocol starting in the early follicular, and luteal menstrual cycle phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early follicular phase protocol (Active Comparator): On day 2 or 3 of the menstrual cycle, following baseline blood sampling, a single SC injection of 150 ìg corifollitropin alfa will be administered (Stimulation Day 1). Starting on Stimulation Day 6, the subject will receive a daily SC injection of 0.25 mg ganirelix up to and including the day of GnRH agonist triggering administration to prevent premature LH surges. From Stimulation Day 8 onwards treatment is continued with a daily SC dose of rFSH (200IU/day) up to the day of GnRHa administration.
  Interventions: Drug: Follicular phase corifollitropin alfa
- Luteal phase protocol (Experimental): Following baseline blood sampling on cycle day 2 of 3 of the menstrual cycle, patients will be followed up with blood and ultrasound from cycle day 10 onwards till the detection of serum LH peak. LH peak will be defined as an increase in serum LH above 20IU/LH. Five (5) days after the LH peak a single SC injection of 150 ìg corifollitropin alfa will be administered (Stimulation Day 1). Starting on Stimulation Day 6, the subject will receive a daily SC injection of 0.25 mg ganirelix up to and including the day of GnRH agonist triggering administration to prevent premature LH surges. From Stimulation Day 8 onwards treatment is continued with a daily SC dose of rFSH (200IU/day) up to the day of GnRHa administration.
  Interventions: Drug: Luteal phase corifollitropin alfa

INTERVENTIONS:
Drug: Follicular phase corifollitropin alfa — GnRH antagonist protocol with corifollitropin alfa initiated in the follicular phase (day 2 or 3 of the menstrual cycle)
  Arms: Early follicular phase protocol
Drug: Luteal phase corifollitropin alfa — GnRH antagonist protocol with corifollitropin alfa initiated in the luteal phase (5 days after an LH peak)
  Arms: Luteal phase protocol

SUMMARY:
To evaluate the effect of random-start of ovarian stimulation initiated in the early follicular or luteal phase on the pharmacokinetics and follicular dynamics and embryo euploidy rates in oocyte donors treated with identical ovarian stimulation protocols with corifollitropin alfa and GnRH antagonist pituitary downregulation

DETAILED DESCRIPTION:
The scope of the current prospective trial is to investigate whether Luteal Stimulation (LS) results in equivalent euploid embryos with Follicular Stimulation (FS) in young reproductive age women. The use of the "oocyte donor model" allows extrapolation of the results and application of LS routinely not only in healthy women undergoing fertility preservation but also in all patients irrespective of the menstrual date. This may indeed allow widespread introduction of LS in IVF programs which may result in proper scheduling of ovarian stimulation which is a major issue in everyday clinical practice.

Given that the pharmacokinetics and follicular dynamics of 150μg corifollitropin alfa for luteal stimulation has never been evaluated, the current study of luteal stimulation with corifollitropin alfa could be very interesting for several reasons:

1. Potentially immediate synchronization of oocyte donors with recipients aiming to fresh oocyte donation.
2. Fertility preservation patients for medical, oncological and non-medical indication
3. Any situation in which endometrial receptivity is not pursued.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy eligible oocyte donors
2. Age 18-34 years
3. AFC >12 and AMH>1.5 ng/ml
4. BMI 19-28kg/m2
5. Body weight >60kg
6. Both ovaries present
7. Willing to participate in the study
8. Willing to use non-hormonal contraception or not needing contraception Recipients will be eligible only if their partners' sperm which will be used for ICSI will be normal. Couples will be excluded in case of moderate to severe oligoasthenospermia.

Exclusion Criteria:

1. Endometriosis
2. AFC>20
3. PCOS
4. Low ovarian reserve
5. Endocrine abnormalities
6. Hormonal contraception
7. Contraindication of hormonal treatment
8. History of Ovarian Hyperstimulation Syndrome or hyper-response (> 30 follicles .

11mm)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Mean number of euploid embryos | 15-45 days following oocyte retrieval procedure
  Number of euploid embryos between oocytes received from follicular phase or luteal phase initiation of ovarian stimulation.

SECONDARY OUTCOMES:
Number of oocytes | 9 -20 days from initiation of ovarian stimulation
  The outcome will be evaluated on the day of oocyte retrieval
Number of MIIs | 9 -20 days from initiation of ovarian stimulation
  The outcome will be evaluated on the day of oocyte retrieval
Total additional dose of rFSH (IU) | 9 -20 days from initiation of ovarian stimulation
  Addition total units of FSH following corifollitropin alfa.The outcome will be evaluated on the day of final oocyte maturation
Duration of ovarian stimulation | 9 -20 days from initiation of ovarian stimulation
  Total days of ovarian stimulation .The outcome will be evaluated on the day of final oocyte maturation
Endocrine profile at specific intervals | Stimulation day 1, day 6, day 8, and Day of final oocyte maturation (actual day may vary between 9-15)
  Estradiol, LH, FSH, Progesterone
Clinical pregnancy rates following transfer of embryos generated from oocytes from follicular phase vs. luteal phase stimulation | 5-8 weeks after embryo transfer procedure
  Clinical pregnancy rates , presence of intrauterine gestational sac with an embryonic pole demonstrating cardiac activity

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Consultorio Dexeus, Barcelona
  - Departamento de Ginecología Obstetricia y Reproducción. Hospital Universitari Dexeus, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Martinez F, Clua E, Roca M, Garcia S, Polyzos NP. Comparison of blastocyst euploidy rates following luteal versus follicular phase stimulation in a GnRH antagonist protocol: a prospective study with repeated ovarian stimulation cycles. Hum Reprod. 2022 Nov 24;37(12):2777-2786. doi: 10.1093/humrep/deac222. PMID 36269092